CLINICAL TRIAL: NCT03138824
Title: Storz Professional Image Enhancement System (SPIES) Versus Conventional White Light Imaging (WLI) Assisted Transurethral Resection of Bladder Tumour (TURBT) for Treatment of Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Storz Professional Image Enhancement System Versus White Light Imaging Assisted TURBT for Treatment of NMIBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Msc, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS/17.03.57
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Bladder Urothelial Carcinoma; TURBT; Bladder Neoplasm; Cystoscopy
Keywords: Bladder Urothelial Carcinoma; TURBT; Recurrence; Progression
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence; Disease Progression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIES assisted TURBT (Experimental): Storz Professional Image Enhancement System (SPIES) assisted transurethral resection of bladder tumour for Non-muscle invasive bladder cancer
  Interventions: Procedure: SPIES assisted TURBT
- WLI assisted TURBT (Experimental): White Light Imaging (WLI) assisted transurethral resection of bladder tumour for Non-muscle invasive bladder cancer
  Interventions: Procedure: WLI assisted TURBT

INTERVENTIONS:
Procedure: SPIES assisted TURBT — SPIES assisted TURBT of NMIBC
  Other Names: Storz Professional Image Enhancement System (SPIES)
  Arms: SPIES assisted TURBT
Procedure: WLI assisted TURBT — White Light Imaging (WLI) assisted TURBT for treatment of NMIBC
  Other Names: White Light Imaging (WLI)
  Arms: WLI assisted TURBT

SUMMARY:
Compare the therapeutic utility of SPIES assisted TURB with WLI assisted TURB in patients with non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
Urothelial carcinoma of the bladder is the 2nd most common urological malignancy. The vast majority of newly diagnosed cases are non-muscle invasive bladder cancers (NMIBC), which represent about 75%, and it can be treated with transurethral resection (TURBT). The goal of TURBT in Ta and T1 NMIBC is to make the correct diagnosis and completely remove all visible lesions. The quality of TURBT strongly determines patient prognosis and overall treatment.

White light cystoscopy (WLC) remains despite of its limitations the cornerstone of the diagnosis and subsequent treatment of NMIBC. The sensitivity and specificity of WLC range from 62% to 84% and 43% to 98%, respectively. Its sensitivity is lower for small papillary bladder tumors and carcinoma in situ (CIS). Moreover, the accuracy of WLC has been shown to be operator dependent.

Smaller or satellite tumors can be missed, which contributes to almost 40% rate of residual bladder cancer found at the time of 'second-look' TUR. Indistinct borders and difficult visualization of submucosal tumor margins during TUR can lead to incomplete tumor resection and understaging of bladder cancer and leads to tumor recurrence which range from 15% to 61% at one year after surgery based on combined analysis of seven EORTC studies. 3 Non-papillary and flat malignant lesions such as carcinoma in situ (CIS) can be difficult to differentiate from inflammation, with detection rates of CIS only 58% to 68% by WLC.

Fluorescence cystoscopy also known as blue light cystoscopy or photodynamic diagnosis (PDD) requires preoperative intravesical administration of protoporphyrin IX precursor as the contrast agent, a blue light source that illuminates at 375 to 440 nm. Protoporphyrin accumulates preferentially in neoplastic cells and emits fluorescence in the red part of the spectrum under blue light excitation. Though PDD also does not distinguish high-grade from low-grade bladder cancer, PDD has an increased rate of detection of flat appearing CIS vs WLC (87% vs 75% pooled sensitivity; P= .006).

The recurrence rate of PDD-guided TUR of bladder tumor is a matter of controversy. In a meta-analysis of prospective studies on 1345 patients with overall 12 months recurrence rate was significantly lower with PDD compared with WLC (34.5% vs 45.4% pooled sensitivity; P=0.006). However, a prospective randomized multi-institutional trial found no difference in tumor recurrence and progression between PDD and WLC.

Narrow band maging (NBI) devices filter out the red spectrum from white light, with the resultant blue (415 nm) and green (540 nm) spectra absorbed by hemoglobin, thus highlighting the contrast between capillaries and mucosa with no significant difference in detection rate of bladder tumor between new and experienced users. Under NBI, the more vascularized CIS or tumor areas are accentuated in appearance as green or brown. However visibility of NBI cystoscopy is reduced with bleeding or inflammation, due to the strong absorption of light by hemoglobin. In contrast to PDD, systems integrating WLC and NBI are already available. In a recent meta-analysis of 8 studies including 1022 patients, the detection of bladder cancer was higher by NBI compared with WLC on a per-person basis (94% vs 85% pooled sensitivity) and a per-lesion basis (95% vs 75% pooled sensitivity); however, the pooled specificity on a per-lesion basis was lower by NBI compared with WLC (55% vs 72%).

Similar to PDD, NBI does not distinguish bladder cancer grade. The detection of CIS was significantly improved by NBI over WLC (100% vs 83% sensitivity) in a study of 427 patients. Another multicenter, prospective study reported a significantly increased sensitivity for the detection of CIS from 50% for WLC to 90% for NBI in 104 patients. In a recent, single-center, randomized, controlled trial to assess whether NBI improved TUR of bladder tumors in 254 patients with 2-year follow-up, a reduced recurrence rate (22% vs 33%; P=.05) and improved recurrence-free survival (22 vs 19 months; P =.02) were reported by NBI compared with WLC.

Storz Professional Image Enhancement System (SPIES) offers several image enhancement modalities: Spectra A mode is based mainly on the green (~500-570 nm) and blue (~400-480 nm) light spectral signals that are separated in the (Red-Green-Blue) of the camera system within these bands the hemoglobin absorption is significantly higher compared to the red spectral band above 570 nm. Due to the limited penetration depth in the blue to green spectral part, this mode allows to highlight the contrast of capillaries and vessels in the superficial mucosa and submucosa. The SPIES Spectra B pronounces as well as the Spectra A mode the blue to green spectral part in order to reach a higher contrast in the superficial mucosa and sub mucosa. However SPECTRA B is obtained by adding 15% of red colour to SPECTRA A. The Chroma modality enhance the sharpness of the image. The Clara modality create a clearer image of darker regions within the image. Together they should provide a clearer and sharper image of the original WL image.

SPIES enhances the blue and the green wavelengths of the transmitted image and a three-colour image is built from these components of the spectral input. This effect is achieved by suppression of the red portion of the spectrum. By adding different colours to the blue- and green-coloured image (e.g. orange or violet), three types of SPIES images are produced, giving the surgeon three different options for visualization. SPIES proposes the option to choose the best enhancement method in different clinical situations, e.g. SPIES A or C mode, if high contrast is desired or SPIES B mode in case of visual interferences during cystoscopy as hematuria.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed at the out-patient cystoscopy with papillary bladder or small resectable lesion that can be resected tumour

Exclusion Criteria:

* Tumor criteria

  a. Beyond scope of resection
* Patients criteria

  1. Poor performance status
  2. History of bladder irradiation
  3. Contracted bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence after TURBT in patients with NMIBC | 3 months after primary procedure
  inpatient cystoscopy of the tumor site for detection of tumor recurrence disease in each arm

SECONDARY OUTCOMES:
1-year recurrence free survival | 1 year
  Number of patients surviving for one year without tumor recurrence will be counted and compared

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mosbah, MD, Phd, Study Chair — Urology and Nephrology Center; Bedir Ali-Eldeen, MD, Phd, Study Director — Urology and Nephrology Center; Ahmed Elshal, MD, Study Director — Urology and Nephrology Center; Abdelwahab Hashem, Msc, Principal Investigator — Urology and Nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Ahmed Elshal, MD